CLINICAL TRIAL: NCT03161314
Title: Plantar Heel Pain: Multisegmental Foot Motion and Muscle Function, FFI Translation, and Evaluation of Physical Therapy Treatments
Brief Title: Plantar Heel Pain: Multisegment Foot Motion and Muscle Function, FFI Translation, and Evaluation of Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Thailand Research Fund (Other)
Responsible Party: Principal Investigator, Sunee Bovonsunthonchai, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MU-CIRB 2016/182.0211
Record Dates: First submitted 2017-05-08; First posted 2017-05-19 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Plantar Fasciitis
Keywords: plantar fasciitis; multisegment foot motion; gait; physical therapy; strengthening; stretching; exercise; translation; plantar heel pain
MeSH Terms: conditions — Fasciitis, Plantar; Motor Activity | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: A stratified randomization table according to age (less or more than 50 years) and pain score (less or more than 5 out of 10 scores) was used.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Conservative physical therapy intervention was launched by the same physical therapist who blind to participant group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strengthening group (Experimental): Individuals with PF who received strengthening exercises. (study 3)
  Interventions: Procedure: Strengthening exercises
- Stretching group (Active Comparator): Individuals with PF who received stretching exercises. (study 3)
  Interventions: Procedure: Stretching exercises

INTERVENTIONS:
Procedure: Strengthening exercises — Conservative physical therapy treatment with home-based strengthening exercises (study 3)
  Arms: Strengthening group
Procedure: Stretching exercises — Conservative physical therapy treatment with home-based stretching exercises (study 3)
  Arms: Stretching group

SUMMARY:
Plantar fasciitis (PF) is a prevalent musculoskeletal condition of plantar heel pain (PHP) that leads to pain, functional limitations, and reduced quality of life, especially among active adults aged 25 to 65. Understanding the biomechanical alterations in foot motion among individuals with PF is essential to inform targeted treatment strategies and prevent symptom chronicity. However, research exploring detailed multi-segment foot motion changes in this population remains limited.

Assessing foot function is a key component in understanding symptom development and treatment outcomes. The Foot Function Index (FFI) is an internationally recognized, reliable, and valid questionnaire used to measure foot pain and disability. To facilitate its use in Thai populations and enable cross-cultural comparisons, it is crucial to translate and validate the FFI into Thai.

Although exercise interventions such as strengthening and stretching are widely used to manage PHP, evidence regarding their relative effectiveness on pain reduction and gait improvement is inconclusive. Rigorous evaluation of these programs is needed to establish evidence-based guidelines for physical therapy in this population.

Study 1: Comparative Study of Gait and Foot Segment Motion Between Individuals with Plantar Fasciitis and Healthy Controls This study aimed to compare multi-segment foot motion during walking between individuals with plantar fasciitis (PF) and healthy controls. A matched case-control design was used, with gait data collected via a 3D motion capture system and analyzed using the Oxford Foot Model.

Study 2: Translation and Validation of the Thai Version of the Foot Function Index (FFI-Th) This study aimed to translate the Foot Function Index (FFI) into Thai (FFI-Th) and evaluate its psychometric properties individuals with plantar foot complaints.

Study 3: Effects of Strengthening and Stretching Exercise Programs on Pain and Gait in Patients with Plantar Fasciitis: A Randomized Controlled Trial This study aimed to investigate the effects of physical therapy interventions-specifically strengthening versus stretching exercise programs-on pain and temporospatial gait parameters in patients with PF.

DETAILED DESCRIPTION:
Procedure

Study 1: Comparative Study of Gait and Foot Segment Motion Between Individuals with Plantar Fasciitis and Healthy Controls

A matched case-control study recruited individuals with PF and matched healthy controls by age, gender, weight, and height. After informed consent, anthropometric data were collected, and participants wore tight clothing to allow accurate marker placement. Forty-two reflective markers were attached to define foot and lower limb segments following the Oxford Foot Model and Plug-In-Gait protocols. A static calibration trial was recorded, after which some markers were removed. Then, participants performed walking trials along an 8-meter walkway while motion capture cameras and force plates recorded kinematic and kinetic data simultaneously. Each participant completed 3-5 gait trials at a self-selected comfortable speed, with two trials matching the control group's gait speed and cadence selected for analysis. Data were filtered and normalized over the gait cycle for further assessment. Outcome measures included ground reaction forces (GRFs) during braking and propulsion phases and peak multi-segment foot joint angles in three planes.

Study 2: Translation and Validation of the Thai Version of the Foot Function Index (FFI-Th)

This study used a cross-sectional design to translate and validate the Foot Function Index (FFI) into Thai (FFI-Th) following a standardized cross-cultural adaptation process. The steps included independent forward translation by two bilingual translators, synthesis by an expert committee, backward translation by two native English speakers, harmonization through consensus meetings, cognitive interviews with 20 individuals to ensure clarity, and final proofreading by a linguist. To assess criterion validity, participants also completed the EuroQol five-dimensional questionnaire (EQ-5D-5L) for health-related quality of life and a pain visual analogue scale (pain-VAS). These instruments provided comparative data for evaluating the FFI-Th's validity.

Study 3; Effects of Strengthening and Stretching Exercise Programs on Pain and Gait in individuals with Plantar Fasciitis: A Randomized Controlled Trial

This double-blind, randomized controlled trial was used. Individuals with PF were screened and recruited based on specific inclusion and exclusion criteria. After obtaining informed consent, participants were randomly assigned into two groups: strengthening exercises or stretching exercises. All participants received a standardized physical therapy treatment including therapeutic ultrasound and manual therapy, followed by their assigned exercise programs instructed by blinded physical therapists. Participants performed home-based exercises three times daily for 4 weeks, then continued at home for 2 months with exercise logs to monitor compliance. Outcome assessments were conducted five times: baseline, mid-intervention, post-intervention, and at 1- and 2-month follow-ups. Data collected included demographics, pain intensity via visual analogue scale (VAS), and temporospatial gait parameters measured by a force distribution platform and synchronized video system.

ELIGIBILITY:
Study 1: Comparative Study of Gait and Foot Segment Motion Between Individuals with Plantar Fasciitis and Healthy Controls

Inclusion Criteria (PF Group):

* Aged 20-80 years
* Plantar fasciitis (PF) symptoms for at least one month
* Pain or tenderness at the medial calcaneal tubercle or proximal plantar fascia
* At least one of the following symptoms:

  * Morning pain (first steps in the morning)
  * Pain after prolonged sitting
  * Pain during weight-bearing activities

Exclusion Criteria (PF Group):

* Other painful conditions in the lower extremity or back
* History of rheumatoid arthritis
* Neurological or vascular diseases
* Leg length discrepancy >1 cm
* Severe pain preventing walking

Inclusion Criteria (Healthy Controls):

* No current or previous history of PF symptoms
* No foot pain

Exclusion Criteria (Healthy Controls):

• Same as those listed for the PF group

Study 2: Translation and Validation of the Thai Version of the Foot Function Index (FFI-Th) Inclusion Criteria (Individuals with plantar problems)

* Aged 20-80 years
* Experienced plantar foot pain or tenderness for at least one month (at rest or during weight-bearing activities)
* Able to read and communicate in Thai
* No uncorrected visual impairments Exclusion Criteria (Individuals with plantar problems)
* Pain in other areas of the lower extremities
* History of systemic inflammatory diseases
* History of neurological diseases
* Received any treatment during the study period

Study 3: Effects of Strengthening and Stretching Exercise Programs on Pain and Gait in Patients with Plantar Fasciitis: A Randomized Controlled Trial Inclusion Criteria:

* Aged 20-80 years
* Heel pain lasting more than one month
* Pain during the first steps in the morning or after rest
* Tenderness at the medial calcaneal tubercle
* Plantar fascia thickness greater than 4.0 mm (confirmed by ultrasound)

Exclusion Criteria:

* History of back or lower limb surgery within 6 months
* Recent trauma or corticosteroid injections (within 6 months)
* Leg length discrepancy greater than 1 cm
* Pregnancy
* Inability to perform the exercise program
* Receiving other ongoing treatments or performing other foot-specific exercises
* Coexisting conditions including:

  * Achilles tendinopathy
  * Acute ankle sprain
  * Tarsal tunnel syndrome
  * Patellofemoral syndrome
  * Calcaneal spurs
  * Heel pad syndrome

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunee Bovonsunthonchai, PhD, Principal Investigator — Mahidol University
Locations (2):
- Thailand (2):
  - Motion analysis laboratory, Salaya, Nakhonpathom
  - Physical therapy center, Physical therapy faculty, Mahidol University, Bangkok

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin RL, Davenport TE, Reischl SF, McPoil TG, Matheson JW, Wukich DK, McDonough CM; American Physical Therapy Association. Heel pain-plantar fasciitis: revision 2014. J Orthop Sports Phys Ther. 2014 Nov;44(11):A1-33. doi: 10.2519/jospt.2014.0303. PMID 25361863
- [Background] Cole C, Seto C, Gazewood J. Plantar fasciitis: evidence-based review of diagnosis and therapy. Am Fam Physician. 2005 Dec 1;72(11):2237-42. PMID 16342847
- [Background] Lemont H, Ammirati KM, Usen N. Plantar fasciitis: a degenerative process (fasciosis) without inflammation. J Am Podiatr Med Assoc. 2003 May-Jun;93(3):234-7. doi: 10.7547/87507315-93-3-234. PMID 12756315
- [Background] Chang R, Rodrigues PA, Van Emmerik RE, Hamill J. Multi-segment foot kinematics and ground reaction forces during gait of individuals with plantar fasciitis. J Biomech. 2014 Aug 22;47(11):2571-7. doi: 10.1016/j.jbiomech.2014.06.003. Epub 2014 Jun 11. PMID 24992816
- [Background] Wearing SC, Smeathers JE, Yates B, Sullivan PM, Urry SR, Dubois P. Sagittal movement of the medial longitudinal arch is unchanged in plantar fasciitis. Med Sci Sports Exerc. 2004 Oct;36(10):1761-7. doi: 10.1249/01.mss.0000142297.10881.11. PMID 15595298
- [Background] Budiman-Mak E, Conrad KJ, Mazza J, Stuck RM. A review of the foot function index and the foot function index - revised. J Foot Ankle Res. 2013 Feb 1;6(1):5. doi: 10.1186/1757-1146-6-5. PMID 23369667
- [Result] Hill CL, Gill TK, Menz HB, Taylor AW. Prevalence and correlates of foot pain in a population-based study: the North West Adelaide health study. J Foot Ankle Res. 2008 Jul 28;1(1):2. doi: 10.1186/1757-1146-1-2. PMID 18822153
- [Result] Sullivan J, Burns J, Adams R, Pappas E, Crosbie J. Musculoskeletal and activity-related factors associated with plantar heel pain. Foot Ankle Int. 2015 Jan;36(1):37-45. doi: 10.1177/1071100714551021. Epub 2014 Sep 18. PMID 25237175
- [Result] Rathleff MS, Moelgaard C, Lykkegaard Olesen J. Intra- and interobserver reliability of quantitative ultrasound measurement of the plantar fascia. J Clin Ultrasound. 2011 Mar-Apr;39(3):128-34. doi: 10.1002/jcu.20787. Epub 2011 Jan 10. PMID 21387326
- [Result] Digiovanni BF, Nawoczenski DA, Malay DP, Graci PA, Williams TT, Wilding GE, Baumhauer JF. Plantar fascia-specific stretching exercise improves outcomes in patients with chronic plantar fasciitis. A prospective clinical trial with two-year follow-up. J Bone Joint Surg Am. 2006 Aug;88(8):1775-81. doi: 10.2106/JBJS.E.01281. PMID 16882901
- [Result] Rathleff MS, Molgaard CM, Fredberg U, Kaalund S, Andersen KB, Jensen TT, Aaskov S, Olesen JL. High-load strength training improves outcome in patients with plantar fasciitis: A randomized controlled trial with 12-month follow-up. Scand J Med Sci Sports. 2015 Jun;25(3):e292-300. doi: 10.1111/sms.12313. Epub 2014 Aug 21. PMID 25145882
- [Derived] Bovonsunthonchai S, Thong-On S, Vachalathiti R, Intiravoranont W, Suwannarat S, Smith R. Thai version of the foot function index: a cross-cultural adaptation with reliability and validity evaluation. BMC Sports Sci Med Rehabil. 2020 Sep 10;12:56. doi: 10.1186/s13102-020-00206-8. eCollection 2020. PMID 32944253

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at Physical Therapy Center, Mahidol University (study 3)
Groups:
- Strengthening Group: Conservative physical therapy with home-based strengthening exercises (study 3)
- Stretching Group: conservative physical therapy with home-based stretching exercises (study 3)
Period: Baseline
Arm/Group | Strengthening Group | Stretching Group
Started | 42 | 42
Completed | 42 | 42
Not Completed | 0 | 0
Period: 2 Weeks After the Intervention
Arm/Group | Strengthening Group | Stretching Group
Started | 42 | 42
Completed | 42 | 42
Not Completed | 0 | 0
Period: 4 Weeks After the Intervention
Arm/Group | Strengthening Group | Stretching Group
Started | 42 | 42
Completed | 42 | 42
Not Completed | 0 | 0
Period: 1-month Follow-up
Arm/Group | Strengthening Group | Stretching Group
Started | 42 | 42
Completed | 42 | 42
Not Completed | 0 | 0
Period: 2-month Follow-up
Arm/Group | Strengthening Group | Stretching Group
Started | 42 | 42
Completed | 42 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Strengthening Group: Conservative physical therapy with home-based strengthening exercises
- Stretching Group: Conservative physical therapy with home-based stretching exercises
- Total: Total of all reporting groups
Arm/Group | Strengthening Group | Stretching Group | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.95 (10.10) | 52.86 (9.84) | 52.40 (9.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 33 | 62
  Male | 13 | 9 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: kg] | 65.66 (11.26) | 65.14 (12.52) | 65.40 (11.90)
Height [Mean (Standard Deviation); unit: cm] | 161.13 (9.18) | 159.45 (8.13) | 160.05 (8.67)
Pain at worst intensity [Mean (Standard Deviation); unit: scores] — Pain at worst intensity was assessed using the Visual analog scale (VAS), where 0 indicates "no pain" and 10 indicates "pain as bad as participants can imagine". Participants were asked to report their worst pain level over the past 24 hours. Higher scores indicate more severe pain. Unit of Measure: scores
  scores | 5.96 (2.3) | 5.74 (2.3) | 5.85 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Worst Pain
Description: Worst pain was assessed using the Visual analog scale (VAS), where 0 indicates "no pain" and 10 indicates "pain as bad as participants can imagine". Participants were asked to report their worst pain level over the past 24 hours. Higher scores indicate more severe pain. Unit of Measure: scores
Time Frame: Baseline, 2 weeks after the intervention, 4 weeks after the intervention, 1-month follow-up, and 2-month follow-up
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Strengthening Group | Stretching Group
Number analyzed (Participants) | 42 | 42
score
  Baseline | 5.96 (2.3) | 5.74 (2.3)
  2 weeks after the intervention | 3.91 (2.38) | 4.08 (2.29)
  4 weeks after the intervention | 3.09 (2.25) | 3.34 (2.47)
  1-month follow-up | 2.52 (2.55) | 2.69 (2.55)
  2-month follow-up | 1.73 (2.16) | 2.69 (2.55)
Statistical Analysis 1: Comparison: Strengthening Group vs Stretching Group; Baseline; Test type: Superiority; p = 0.660, t-test, 2 sided
Statistical Analysis 2: Comparison: Strengthening Group vs Stretching Group; 2 weeks after the intervention; Test type: Superiority; p = 0.734, t-test, 2 sided
Statistical Analysis 3: Comparison: Strengthening Group vs Stretching Group; 4 weeks after the intervention; Test type: Superiority; p = 0.629, t-test, 2 sided
Statistical Analysis 4: Comparison: Strengthening Group vs Stretching Group; 1-month follow-up; Test type: Superiority; p = 0.752, t-test, 2 sided
Statistical Analysis 5: Comparison: Strengthening Group vs Stretching Group; 2-month follow-up; Test type: Superiority; p = 0.512, t-test, 2 sided
Statistical Analysis 6: Comparison: Strengthening Group; Within group comparison; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 7: Comparison: Stretching Group; Within group comparison; Test type: Superiority; p < 0.001, ANOVA

2. Primary Outcome: Morning Pain
Description: Morning pain intensity upon waking was assessed using a 10 cm Visual Analog Scale (VAS), where participants mark a point along a continuous line anchored by "no pain" (0) and "worst imaginable pain" (10), with higher values indicating more severe morning pain. Unit of Measure: scores
Time Frame: Baseline, 2 weeks after the intervention, 4 weeks after the intervention, 1-month follow-up, and 2-month follow-up
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Strengthening Group | Stretching Group
Number analyzed (Participants) | 42 | 42
score
  Baseline | 5.86 (2.51) | 5.04 (2.35)
  2 weeks after the intervention | 3.70 (2.28) | 3.63 (2.54)
  4 weeks after the intervention | 2.90 (2.46) | 2.75 (2.52)
  1-month follow-up | 2.25 (2.51) | 1.98 (2.24)
  2-month follow-up | 1.30 (1.54) | 1.52 (2.12)
Statistical Analysis 1: Comparison: Strengthening Group vs Stretching Group; Baseline; Test type: Superiority; p = 0.128, t-test, 2 sided
Statistical Analysis 2: Comparison: Strengthening Group vs Stretching Group; 2 weeks after the intervention; Test type: Superiority; p = 0.889, t-test, 2 sided
Statistical Analysis 3: Comparison: Strengthening Group vs Stretching Group; 4 weeks after the intervention; Test type: Superiority; p = 0.793, t-test, 2 sided
Statistical Analysis 4: Comparison: Strengthening Group vs Stretching Group; 1-month follow-up; Test type: Superiority; p = 0.602, t-test, 2 sided
Statistical Analysis 5: Comparison: Strengthening Group vs Stretching Group; 2-month follow-up; Test type: Superiority; p = 0.574, t-test, 2 sided
Statistical Analysis 6: Comparison: Strengthening Group; Within group comparison; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 7: Comparison: Stretching Group; Within group comparison; Test type: Superiority; p < 0.001, ANOVA

3. Secondary Outcome: Cadence
Description: Cadence refers to the number of steps taken per minute during walking. It is a critical parameter in gait analysis, influencing both performance and injury risk, and the effectiveness of rehabilitation programs. Unit of Measure: steps/minute
Time Frame: Baseline, 2 weeks after the intervention, 4 weeks after the intervention, 1-month follow-up, and 2-month follow-up
Measure: Mean (Standard Deviation); unit: steps/minute
Arm/Group | Strengthening Group | Stretching Group
Number analyzed (Participants) | 42 | 42
steps/minute
  Baseline | 103.16 (7.75) | 101.37 (10.44)
  2 weeks after the intervention | 102.85 (8.54) | 103.70 (9.82)
  4 weeks after the intervention | 104.03 (8.42) | 103.46 (10.42)
  1-month follow-up | 104.72 (8.45) | 104.16 (9.35)
  2-month follow-up | 105.50 (8.47) | 104.81 (9.49)
Statistical Analysis 1: Comparison: Strengthening Group vs Stretching Group; Baseline; Test type: Superiority; p = 0.374, t-test, 2 sided
Statistical Analysis 2: Comparison: Strengthening Group vs Stretching Group; 2 weeks after the intervention; Test type: Superiority; p = 0.674, t-test, 2 sided
Statistical Analysis 3: Comparison: Strengthening Group vs Stretching Group; 4 weeks after the intervention; Test type: Superiority; p = 0.781, t-test, 2 sided
Statistical Analysis 4: Comparison: Strengthening Group vs Stretching Group; 1-month follow-up; Test type: Superiority; p = 0.778, t-test, 2 sided
Statistical Analysis 5: Comparison: Strengthening Group vs Stretching Group; 2-month follow-up; Test type: Superiority; p = 0.727, t-test, 2 sided
Statistical Analysis 6: Comparison: Strengthening Group; Within group comparison; Test type: Superiority; p = 0.014, ANOVA
Statistical Analysis 7: Comparison: Stretching Group; Within group comparison; Test type: Superiority; p = 0.002, ANOVA

4. Secondary Outcome: Stride Length
Description: Stride length is the distance covered between two consecutive placements of the same foot during walking. It represents the length of a full gait cycle, encompassing both the stance and swing phases of the same limb. In clinical assessments, stride length is measured to evaluate gait efficiency, balance, and the effectiveness of rehabilitation program. Unit of Measure: meter
Time Frame: Baseline, 2 weeks after the intervention, 4 weeks after the intervention, 1-month follow-up, and 2-month follow-up
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Strengthening Group | Stretching Group
Number analyzed (Participants) | 42 | 42
meter
  Baseline | 1.05 (0.11) | 1.03 (0.10)
  2 weeks after the intervention | 1.06 (0.10) | 1.06 (0.10)
  4 weeks after the intervention | 1.05 (0.10) | 1.05 (0.10)
  1-month follow-up | 1.07 (0.09) | 1.07 (0.11)
  2-month follow-up | 1.07 (0.10) | 1.08 (0.10)
Statistical Analysis 1: Comparison: Strengthening Group vs Stretching Group; Baseline; Test type: Superiority; p = 0.390, t-test, 2 sided
Statistical Analysis 2: Comparison: Strengthening Group vs Stretching Group; 2 weeks after the intervention; Test type: Superiority; p = 0.770, t-test, 2 sided
Statistical Analysis 3: Comparison: Strengthening Group vs Stretching Group; 4 weeks after the intervention; Test type: Superiority; p = 0.603, t-test, 2 sided
Statistical Analysis 4: Comparison: Strengthening Group vs Stretching Group; 1-month follow-up; Test type: Superiority; p = 0.922, t-test, 2 sided
Statistical Analysis 5: Comparison: Strengthening Group vs Stretching Group; 2-month follow-up; Test type: Superiority; p = 0.560, t-test, 2 sided
Statistical Analysis 6: Comparison: Strengthening Group; Within group comparison; Test type: Superiority; p = 0.181, ANOVA
Statistical Analysis 7: Comparison: Stretching Group; Within group comparison; Test type: Superiority; p < 0.001, ANOVA

5. Secondary Outcome: Stride Time
Description: Time spend during walking over one gait cycle (s)
  Stride time refers to the duration of one full gait cycle, measured from the initial contact of one foot to the subsequent initial contact of the same foot. It encompasses both the stance and swing phases of the limb's movement. Stride time is a critical temporal parameter in gait analysis, providing insights into the rhythm and coordination of walking. Unit of Measure: second
Time Frame: Baseline, 2 weeks after the intervention, 4 weeks after the intervention, 1-month follow-up, and 2-month follow-up
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Strengthening Group | Stretching Group
Number analyzed (Participants) | 42 | 42
second
  Baseline | 1.17 (0.09) | 1.19 (0.13)
  2 weeks after the intervention | 1.17 (0.10) | 1.16 (0.12)
  4 weeks after the intervention | 1.15 (0.10) | 1.17 (0.13)
  1-month follow-up | 1.15 (0.10) | 1.16 (0.11)
  2-month follow-up | 1.14 (0.10) | 1.15 (0.11)
Statistical Analysis 1: Comparison: Strengthening Group vs Stretching Group; Baseline; Test type: Superiority; p = 0.334, t-test, 2 sided
Statistical Analysis 2: Comparison: Strengthening Group vs Stretching Group; 2 weeks after the intervention; Test type: Superiority; p = 0.766, t-test, 2 sided
Statistical Analysis 3: Comparison: Strengthening Group vs Stretching Group; 4 weeks after the intervention; Test type: Superiority; p = 0.598, t-test, 2 sided
Statistical Analysis 4: Comparison: Strengthening Group vs Stretching Group; 1-month follow-up; Test type: Superiority; p = 0.682, t-test, 2 sided
Statistical Analysis 5: Comparison: Strengthening Group vs Stretching Group; 2-month follow-up; Test type: Superiority; p = 0.707, t-test, 2 sided
Statistical Analysis 6: Comparison: Strengthening Group; Within group comparison; Test type: Superiority; p = 0.008, ANOVA
Statistical Analysis 7: Comparison: Stretching Group; Within group comparison; Test type: Superiority; p = 0.002, ANOVA

6. Secondary Outcome: Gait Speed
Description: Distance of walking over time (m/s)
  Gait speed refers to the rate at which an individual walks. It serves as a crucial indicator of mobility and overall physical fitness, playing a significant role in assessing an individual's balance, endurance, and functional abilities. Unit of Measure: meter/second
Time Frame: Baseline, 2 weeks after the intervention, 4 weeks after the intervention, 1-month follow-up, and 2-month follow-up
Measure: Mean (Standard Deviation); unit: meter/second
Arm/Group | Strengthening Group | Stretching Group
Number analyzed (Participants) | 42 | 42
meter/second
  Baseline | 0.90 (0.11) | 0.87 (0.13)
  2 weeks after the intervention | 0.91 (0.12) | 0.91 (0.13)
  4 weeks after the intervention | 0.92 (0.12) | 0.91 (0.13)
  1-month follow-up | 0.93 (0.12) | 0.93 (0.13)
  2-month follow-up | 0.94 (0.12) | 0.94 (0.13)
Statistical Analysis 1: Comparison: Strengthening Group vs Stretching Group; Baseline; Test type: Superiority; p = 0.287, t-test, 2 sided
Statistical Analysis 2: Comparison: Strengthening Group vs Stretching Group; 2 weeks after the intervention; Test type: Superiority; p = 0.861, t-test, 2 sided
Statistical Analysis 3: Comparison: Strengthening Group vs Stretching Group; 4 weeks after the intervention; Test type: Superiority; p = 0.641, t-test, 2 sided
Statistical Analysis 4: Comparison: Strengthening Group vs Stretching Group; 1-month follow-up; Test type: Superiority; p = 0.864, t-test, 2 sided
Statistical Analysis 5: Comparison: Strengthening Group vs Stretching Group; 2-month follow-up; Test type: Superiority; p = 0.888, t-test, 2 sided
Statistical Analysis 6: Comparison: Strengthening Group; Within group comparison; Test type: Superiority; p = 0.262, ANOVA
Statistical Analysis 7: Comparison: Stretching Group; Within group comparison; Test type: Superiority; p < 0.001, ANOVA

ADVERSE EVENTS:
Time Frame: 3 months in total per participants. Adverse events were monitored over a total of 3 months, which includes a 4-week (1-month) intervention phase plus a subsequent 2-month follow-up phase.
Arm/Group | Strengthening Group | Stretching Group
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

LIMITATIONS AND CAVEATS:
This study did not compare to the pure conservative physical therapy treatment, which may provide more information about the effectiveness of strengthening and stretching exercises that may superior to the conservative treatment alone.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT03161314/Prot_SAP_000.pdf